CLINICAL TRIAL: NCT01550588
Title: Device Closure Versus Medical Therapy for Secondary Prevention in Cryptogenic Stroke Patients With High-Risk Patent Foramen Ovale : DEFENSE-PFO
Brief Title: Device Closure Versus Medical Therapy for Cryptogenic Stroke Patients With High-Risk Patent Foramen Ovale (DEFENSE-PFO)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jae-Kwan Song (Other)
Responsible Party: Sponsor-Investigator, Jae-Kwan Song, professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-0553
Record Dates: First submitted 2012-02-26; First posted 2012-03-12 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Patent Foramen Ovale
Keywords: PFO; Stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke | interventions — Vascular Closure Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medication (Placebo Comparator): Anticoagulation, Antiplatelet agent
  Interventions: Drug: Standard medical treatment
- Device closure (Active Comparator): Amplatzer PFO occluder device
  Interventions: Device: Device closure

INTERVENTIONS:
Device: Device closure — PFO Amplatzer device closure
  Other Names: PFO Amplatzer device
  Arms: Device closure
Drug: Standard medical treatment — Standard Medical management using anti-coagulant therapy
  Arms: Medication

SUMMARY:
Background and hypothesis:

The appropriate treatment strategy for secondary stroke prevention in patients with cryptogenic stroke and patent foramen ovale (PFO) remains challenging. Clinical and anatomical variables reported to be risk factors associated with stroke recurrence include older age, large PFO, large right-to-left shunting, and combined atrial septal aneurysm (ASA), which, however, were not confirmed by other studies. The investigators hypothesized that percutaneous closure of PFO could be an effective option for secondary prevention in cryptogenic stroke patients with high-risk PFO.

Trial Objective:

The primary objective of this study is to assess whether percutaneous device closure of PFO is superior to conventional antithrombotic treatment in preventing stroke recurrence in the cryptogenic stroke patients with high-risk PFO.

DETAILED DESCRIPTION:
Selection of patients:

Among cryptogenic stroke patients, patients who was identified as high risk PFO which might be defined as high-risk of recurrence (PFO size ≥ 2 mm or atrial septal aneurysm or hypermobility by TEE) will be randomized 1:1 to :a) Device closure using Amplatzer device vs. b) standard medical therapy alone. All patients will be followed for at least 2 years.

Echocardiography Findings for high-risk PFO Digitally, stored transesophageal echocardiographic images were reviewed and analyzed by an investigator. Using calipers, the PFO size was measured as the maximum separation of the septum primum from the septum secundum. ASA or hypermobility was defined as ≥ 10 mm of phasic septal excursion either into the atrium or a sum total excursion of ≥ 15 mm during the cardiorespiratory cycle, with a base of ≥ 15 mm.

Web-based 1:1 blinded randomization for

* Experimental Percutaneous Device Closure using AMPLATZER PFO Occluder
* Active Comparator Standard Medical management using anti-coagulant therapy (at least 3 or 6 months) Study Endpoints
* Primary outcome

  * Recurrence of nonfatal stroke/vascular death/TIMI-major bleeding
* Secondary outcome

  * Recurrent nonfatal stroke
  * Vascular death
  * Major bleeding associated with medication
  * Asymptomatic recurrent ischemic stroke on follow-up MR
  * Complete closure of the defect demonstrated by TEE and bubble study (device group) Frequency of residual shunt, (in)correct device position, need for implantation of second device and peri-procedural complications
  * Procedure related complications
  * Medication related complications

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had a cryptogenic stroke within the previous 3 months, radiologically verified
* Subjects who have been diagnosed with a high-risk* Patent Foramen Ovale (PFO), echocardiographically verified (*PFO size ≥ 2 mm or atrial septal aneurysm or hypermobility by TEE)
* Subjects willing to participate in follow-up visits
* Absence of other potential causes of stroke

Exclusion Criteria:

* Any identifiable cause of thromboembolic cause other than PFO
* Subjects with intracardiac thrombus or tumor, dilated cardiomyopathy, prosthetic heart valve or mitral stenosis, endocarditis
* Subjects with significant atherosclerosis or dissection of the aorta, collagen vascular disease, arteritis, vasculitis and coagulopathy
* Subjects who have an acute or recent (within 6 months) myocardial infarction or unstable angina
* Subjects who have a non-vascular origin of the neurological symptoms after brain imaging (CT scan or MRI)
* History of intracranial bleeding, confirmed arterio-venous malformation,aneurysm or uncontrolled coagulopathy
* Pre-existing neurological disorders or intracranial disease, e.g. multiple sclerosis
* Subjects with left ventricular aneurysm or akinesis
* Subjects with atrial fibrillation/atrial flutter (chronic or intermittent)
* Subjects with another source of right to left shunt identified at baseline, including an atrial septal defect and/or fenestrated septum
* Subjects who could not undergo the TEE examination
* Subjects with contraindication to aspirin or Clopidogrel therapy
* Pregnant or desire to become pregnant within the next year
* Subjects who have a underlying malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2012-02; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence of nonfatal stroke / vascular death / TIMI-major bleeding | 2-year

SECONDARY OUTCOMES:
Recurrent nonfatal stroke | 2-year
Vascular death | 2-year
Major bleeding associated with medication | 2-year
Asymptomatic recurrent ischemic stroke on follow-up MR | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Kwan Song, MD, PhD, Principal Investigator — Department of medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (4):
- South Korea (4):
  - YangSan Busan University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Gang Neung Asan Hospital, Gangneung
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Turc G, Lee JY, Brochet E, Kim JS, Song JK, Mas JL; CLOSE and DEFENSE-PFO Trial Investigators. Atrial Septal Aneurysm, Shunt Size, and Recurrent Stroke Risk in Patients With Patent Foramen Ovale. J Am Coll Cardiol. 2020 May 12;75(18):2312-2320. doi: 10.1016/j.jacc.2020.02.068. PMID 32381162
- [Derived] Lee PH, Song JK, Kim JS, Heo R, Lee S, Kim DH, Song JM, Kang DH, Kwon SU, Kang DW, Lee D, Kwon HS, Yun SC, Sun BJ, Park JH, Lee JH, Jeong HS, Song HJ, Kim J, Park SJ. Cryptogenic Stroke and High-Risk Patent Foramen Ovale: The DEFENSE-PFO Trial. J Am Coll Cardiol. 2018 May 22;71(20):2335-2342. doi: 10.1016/j.jacc.2018.02.046. Epub 2018 Mar 12. PMID 29544871